CLINICAL TRIAL: NCT01367535
Title: A Phase I, Randomized, Open-Label, Active- and Placebo-Controlled Parallel Group Study of the Effect of Subcutaneous and Intravenous Methylnaltrexone on CYP450 2D6 Activity in Healthy Extensive Metabolizers of Dextromethorphan
Brief Title: Effects of MNTX on CYP450 2D6 in Metabolizers of Dextromethorphan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Tage Ramakrishna, M.D.;, Progenics Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MNTX 1108
Record Dates: First submitted 2011-05-27; First posted 2011-06-07 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Healthy Adults
MeSH Terms: interventions — methylnaltrexone; Paroxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Experimental)
  Interventions: Drug: SC Methylnaltrexone (MNTX)
- Arm 2 (Experimental)
  Interventions: Drug: IV Methylnaltrexone (MNTX)
- Arm 3 (Active Comparator)
  Interventions: Drug: Oral Paroxetine
- Arm 4 (Placebo Comparator)
  Interventions: Drug: SC Placebo

INTERVENTIONS:
Drug: SC Methylnaltrexone (MNTX)
  Arms: Arm 1
Drug: IV Methylnaltrexone (MNTX)
  Arms: Arm 2
Drug: Oral Paroxetine
  Arms: Arm 3
Drug: SC Placebo
  Arms: Arm 4

SUMMARY:
This study is a single-center, randomized, open-label, active and placebo-controlled, parallel-group, conducted in healthy male volunteers who have been shown to be extensive metabolizers of dextromethorphan.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males between the ages of 18 and 55
2. Non-Smokers
3. Body weight range form 154-220 lbs
4. No history of clinically significant metabolic disorders.

Exclusion Criteria:

1. Any history of low CYP450 2D6 activity
2. History of alcohol abuse or recreational drugs
3. History of any clinically significant disease or condition affecting a major organ system
4. Donation or loss of blood, 60 days proceeding to screening visit.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2006-03; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Plasma Concentration of MNTX | 4 months
  The objective of this study is to assess the effect of SC or IV doses of MNTX on CYP450 2D6 activity.

SECONDARY OUTCOMES:
Plasma Concentration of Paroxetine | 4 months
  The objective of this study is to assess the effect of SC or IV doses of MNTX on CYP450 2D6 activity.

CONTACTS AND LOCATIONS:
Overall Officials: Tage Ramakrishna, MD, Study Director — Progenics Pharmaceuticals, Inc.
Locations (1):
- Progenics Pharmaceuticals, Tarrytown, New York, United States